CLINICAL TRIAL: NCT01980589
Title: A Multicenter, Open-label, Phase 1b Study of Carfilzomib, Cyclophosphamide and Dexamethasone in Newly Diagnosed Multiple Myeloma Subjects
Acronym: CHAMPION 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; WW Domain-Containing Oxidoreductase; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib, Cyclophosphamide and Dexamethasone (CCd) (Experimental): Participants received carfilzomib, cyclophosphamide and dexamethasone for up to eight 28-day cycles, or until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib administered as a 30-minute intravenous (IV) infusion on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. On Days 1 and 2 of Cycle 1, all participants received carfilzomib at 20 mg/m².
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
Drug: Cyclophosphamide — Cyclophosphamide administered orally (PO) at the dose of 300 mg/m² on Days 1, 8, and 15 of each 28-day cycle.
Drug: Dexamethasone — Dexamethasone administered PO or IV at 40 mg on Days 1, 8, 15, and 22 of each 28-day cycle.

SUMMARY:
The primary objective was to determine the maximum tolerated dose of carfilzomib given twice weekly in combination with cyclophosphamide and dexamethasone for patients with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma
2. Measurable disease, as defined by 1 or more of the following

   * Serum M-protein ≥ 0.5 g/dL, or
   * Urine M-protein ≥ 200 mg/24 hours, or
   * In subjects without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal kappa lambda ( κ/λ) ratio
3. Males and females ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Adequate hepatic function
6. Left ventricular ejection fraction (LVEF) ≥ 40%
7. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
8. Platelet count ≥ 50 × 10^9/L
9. Calculated or measured creatinine clearance (CrCl) of ≥ 15 mL/min

Exclusion Criteria:

1. Planned autologous hematopoietic stem cell transplantation (HSCT) for the initial therapy of newly diagnosed multiple myeloma
2. Multiple myeloma of immunoglobulin M (IgM) subtype
3. Prior systemic treatment for multiple myeloma
4. Glucocorticoid therapy within 14 days prior to enrollment that equals or exceeds the equivalent of dexamethasone 160 mg
5. Known amyloidosis
6. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 6 months prior to enrollment.
7. Known human immunodeficiency virus (HIV) seropositive, hepatitis C infection, and/or hepatitis B (subjects with hepatitis B surface antigen [SAg] or core antibody receiving and responding to antiviral therapy directed at hepatitis B are allowed)
8. Significant neuropathy (Grades ≥ 2) within 14 days prior to enrollment
9. Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- United States (9):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - James R. Berenson, MD, West Hollywood, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Horizon Oncology Research, Lafayette, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Clinical Research Alliance, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 centers in the United States.
Pre-assignment Details: Eligible participants were enrolled into sequential dose-escalation cohorts consisting of 3 to 6 participants to establish the maximum tolerated dose (MTD) of carfilzomib when given in combination with cyclophosphamide and dexamethasone. Additional participants were enrolled in an expansion cohort at the established MTD to collect safety data.
Groups:
- Carfilzomib 36 mg/m²: Participants received 36 mg/m² carfilzomib IV infusion on days 1, 2, 8, 9,15, and 16 of each 28 day cycle (on days 1 and 2 of cycle 1, all participants received carfilzomib at 20 mg/m²), cyclophosphamide administered orally at 300 mg/m² on days 1, 8, and 15, and 40 mg dexamethasone on days 1, 8, 15, and 22, for up to eight 28 day cycles, or until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
- Carfilzomib 45 mg/m²: Participants received 45 mg/m² carfilzomib IV infusion on days 1, 2, 8, 9,15, and 16 of each 28 day cycle (on days 1 and 2 of cycle 1, all participants received carfilzomib at 20 mg/m²), cyclophosphamide administered orally at 300 mg/m² on days 1, 8, and 15, and 40 mg dexamethasone on days 1, 8, 15, and 22, for up to eight 28 day cycles, or until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
- Carfilzomib 56 mg/m²: Participants received 56 mg/m² carfilzomib IV infusion on days 1, 2, 8, 9,15, and 16 of each 28 day cycle (on days 1 and 2 of cycle 1, all participants received carfilzomib at 20 mg/m²), cyclophosphamide administered orally at 300 mg/m² on days 1, 8, and 15, and 40 mg dexamethasone on days 1, 8, 15, and 22, for up to eight 28 day cycles, or until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Started | 3 | 3 | 16
Completed | 3 | 3 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m² | Total
Number analyzed (Participants) | 3 | 3 | 16 | 22
Age, Continuous [Median (Full Range); unit: years] | 56.0 [53 to 71] | 63.0 [61 to 66] | 65.0 [49 to 81] | 62.5 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 7 | 9
  Male | 3 | 1 | 9 | 13
Race [Number; unit: participants]
  Asian | 1 | 0 | 1 | 2
  Black or African American | 1 | 1 | 3 | 5
  White | 1 | 2 | 11 | 14
  Other | 0 | 0 | 1 | 1
European Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 1 | 1 | 7 | 9
    1 (Restrictive but ambulatory) | 2 | 2 | 8 | 12
    2 (Ambulatory but unable to work) | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The MTD is defined as the highest carfilzomib dose at which fewer than 33% of participants experience a treatment-related dose-limiting toxicity (DLT) during the first 28-day cycle. The number of participants who experienced a DLT is reported.
  Dose-limiting toxicities are defined as any of the following carfilzomib-related adverse events:
  Nonhematologic:
  * ≥ Grade 3 non-hematological toxicity
  * ≥ Grade 3 acute kidney injury (creatinine > 3 × baseline or > 4.0 mg/dL) lasting > 72 hours
  Hematologic:
  * Grade 4 neutropenia (absolute neutrophil count [ANC] < 0.5 × 10^9/L) lasting for > 7 days
  * Febrile neutropenia (ANC < 1.0 × 10^9/L with a fever ≥ 38.3ºC) of any duration
  * Grade 4 thrombocytopenia (< 25 × 10^9/L) that persists for > 14 days, despite holding treatment
  * Grade 3 or 4 thrombocytopenia associated with > Grade 1 bleeding
Time Frame: First cycle treatment over 28-days
Population: The Safety population is defined as all enrolled participants who received any study treatment.
Measure: Number; unit: participants
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Number analyzed (Participants) | 3 | 3 | 16
participants | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Participants were evaluated for disease response and progression by the investigator according to the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC). Disease response and progression assessments included serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), serum immunofixation, serum free light chain (SFLC), bone marrow sample (including fluorescent in situ hybridization [FISH]), plasmacytoma evaluation, and skeletal survey. Overall response rate is defined as the percentage of participants with a best response of stringent complete response, complete response, very good partial response (VGPR), or partial response.
Time Frame: Disease response was assessed at the end of each cycle and 30 days after the last treatment; maximum treatment duration was 32 weeks.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Number analyzed (Participants) | 3 | 3 | 16
percentage of participants | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 87.5 [61.7 to 98.4]

3. Secondary Outcome: Time To Response (TTR)
Description: Time to response is defined as months from treatment start to first documentation of response of partial response or better. Summary of time to response includes confirmed responders of PR or better only.
Time Frame: as for outcome 2
Population: Participants with an overall response
Measure: Median (Full Range); unit: months
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Number analyzed (Participants) | 2 | 3 | 14
months | 1.3 [1.0 to 1.6] | 0.8 [0.7 to 1.9] | 1.0 [0.9 to 2.8]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 and using the following scale:
  Grade 1 = Mild, Grade 3 = Moderate; Grade 3 = Severe, Grade 4 = Life-threatening; Grade 5 = Fatal.
Time Frame: From first dose of study drug until 30 days after last dose; median duration of treatment was 31 weeks.
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Number analyzed (Participants) | 3 | 3 | 16
participants
  Any adverse event | 3 | 3 | 16
  Adverse event ≥ Grade 3 | 3 | 3 | 10
  Serious adverse events | 0 | 1 | 5
  AE leading to discontinuation of study drug | 0 | 1 | 4
  Fatal adverse events | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 30 days after the last dose; median duration of treatment was 31 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Carfilzomib 36 mg/m² | Carfilzomib 45 mg/m² | Carfilzomib 56 mg/m²
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 5/16
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib 36 mg/m² (N=3) | Carfilzomib 45 mg/m² (N=3) | Carfilzomib 56 mg/m² (N=16)
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib 36 mg/m² (N=3) | Carfilzomib 45 mg/m² (N=3) | Carfilzomib 56 mg/m² (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 9
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 11
Vomiting (Gastrointestinal disorders) | 1 | 2 | 6
Application site rash (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2
Breakthrough pain (General disorders) | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 1
Catheter site pruritus (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 1 | 3
Fatigue (General disorders) | 1 | 0 | 8
Feeling abnormal (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Mass (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 5
Pain (General disorders) | 0 | 1 | 3
Peripheral swelling (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 5
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 5
Blood iron decreased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Urine output increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 3
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5
Ageusia (Nervous system disorders) | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 6
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 2
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Testicular mass (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Interstitial granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 2 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.